CLINICAL TRIAL: NCT00877838
Title: A Phase 2a Study of the Safety and Effectiveness of NXN-188 for the Acute Treatment of Migraine Attacks With Aura
Brief Title: Study of the Safety and Effectiveness of NXN-188 for the Acute Treatment of Migraine Attacks With Aura
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Collaborators: NeurAxon Inc. (Industry)
Responsible Party: Peer Tfelt-Hansen MD., Dr. Med. Sci., Department of Neurology, Glostrup Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NXN-188-202
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Migraine With Aura
Keywords: Headache; Migraine; Aura; Acute; Attack; Clinical; Trial; Intervention; Nitrogen Oxide; NOS; nNOS; Triptan; 5HT; Serotonin
MeSH Terms: conditions — Migraine with Aura; Headache; Migraine Disorders; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NXN-188 — NXN-188 600 mg (3 gelatin capsules each containing 200 mg) when experiencing migraine aura.
Drug: Placebo — Gelatin capsules resembling the ones containing the active substance

SUMMARY:
The following study is being conducted to explore the safety and effectiveness of a new chemical entity called NXN-188 in subjects with a history of migraine with aura. In this study subjects will treat two attacks of migraine with aura during the aura phase - once with placebo and once with NXN-188.

DETAILED DESCRIPTION:
The purpose of this study is to examine a new chemical entity with 5HT agonist activity and an inhibition of the nitric oxide synthase enzyme (NOS) in patients suffering from migraine with aura. Nitric oxide has diverse roles both in normal and pathological processes including the regulation of blood pressure, neurotransmission, and macrophage defense systems. NO is synthesized by three isoforms of the NOS enzyme: neuronal (n), inducible (i) and endothelial (e). Neuronal NOS (nNOS) is found mainly in neuronal tissue and regulates changes in response sensitivity and cellular plasticity; iNOS is found in macrophages and other tissue, produces NO in response to stress and injury and is one source of inflammation; eNOS is found in endothelial cells, responsible for vascular homeostasis and the presumed mechanism for the effects of nitroglycerine therapy in angina; nitroglycerine is an NO donor. NXN-188 is selectively inhibits nNOS.

There is ample scientific and clinical evidence that NO is involved in the pathogenesis of migraine pain, as well as other pain states characterized by central sensitization (e.g., neuropathic pain). NO donors such as trinitroglycerine induce headache followed by migraine in migraineurs with or without aura ; moreover, platelet nitrates (a signal for increased NO) increase before and during a migraine attack. In addition, increasing NO levels can enhance pain responses in animals, including allodynia in rats; NO is a component of several pathways where pain systems converge in the PNS and CNS and regulates the activity of numerous transmitter systems ; NO is involved in central sensitization particularly those involving NMDA and calcium channels and thought to be a major component of the formation of neuropathic pain states Non-specific NOS inhibitors have been reported to relieve migraine and chronic tension type headaches in human studies. In animals, NOS inhibitors reduce pain-related behaviors in multiple neuropathic pain models and spinal cord ischemia as well as reducing pain related behaviors in chemically-induced pain models, particularly in secondary pain states.

The development of central sensitization in the course of a migraine attack suggests a role for the neuronal isoform of the NOS enzyme.

NXN-188 can bind to both 5-HT1D and 5-HT1B receptors with potency similar to sumatriptan; it also selectively binds to nNOS with a level of nNOS inhibition similar to L-NMMA. NXN-188 is devoid of any relevant eNOS inhibition in in vitro cloned human enzyme assays or ex vivo in human coronary arteries and is expected to be effective in treating migraine by inhibition of the nNOS enzyme without vasoconstrictive effects associated with non-selective compounds such as L-NMMA.

The following study is being conducted to further explore NXN-188 response in subjects with a migraine history of aura. In this study subjects will treat two attacks of migraine with aura during the aura phase - once with placebo and once with NXN-188.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female migraineurs with aura between 18 and 65 years old, inclusive
2. Meets the following criteria for migraine headache with aura:

   * Diagnosed with a history of migraine with aura
   * Aura consisting of at least one of the following, but no muscle weakness or paralysis:

     * Fully reversible visual symptoms (e.g. flickering lights, spots, lines, loss of vision)
     * Fully reversible sensory symptoms (e.g. pins and needles, numbness)
     * Fully reversible dysphasia (speech disturbance)
   * Aura has at least two of the following characteristics:

     * Visual symptoms affecting just one side of the field of vision and/or sensory symptoms affecting just one side of the body
     * At least one aura symptom develops gradually over more than 5 minutes and/or different aura symptoms occur one after the other over more than 5 minutes
     * Each symptom lasts from 5-60 minutes
3. At least one migraine headache with aura every 8-weeks and resulting in moderate to severe pain (on a 4-point categorical scale) within 2 hours of the onset of aura.
4. Migraine pain following aura in at least 75% of occurrences
5. The subject has a body mass index (BMI) within the range of 18 to 32
6. The subject is in general good health as determined by the medical history, physical exam, clinical laboratory tests, vital signs [heart rate (HR) and blood pressure (BP; after a 3-minute sitting period)] and ECG

   • ALT cannot be above 1.5x upper limit of normal; creatinine and urea must be within normal limits
7. The subject must be able to speak, read, and understand Danish sufficiently to understand the nature of the study, to provide written informed consent, and complete all study assessments
8. The subject is willing and able to comply with all testing requirements defined in the protocol
9. All females will avoid pregnancy at least 10 days before Visit 1, during the study and up until 3 months after Visit 2
10. Women of childbearing potential must be using a reliable form of contraception. A reliable form of contraception is defined as follows:

    * sterilisation (via hysterectomy or bilateral tubal ligation)
    * sterilisation of partner
    * IUD,
    * birth control pills on stable dose for at least three months before Visit 1, and one month after visit 2.
    * Medroxyprogesterone acetate (Depo-Provera) or etonogestrel (implanon) active for at least three months prior to the study and with continued administration at intervals sufficient to maintain contraceptive efficacy throughout the study period and at least one month after visit 2. Males must use condoms as contraception.

Exclusion Criteria:

1. Presence of any clinically significant condition that would preclude study participation, as evaluated by the investigator
2. Are pregnant or lactating
3. History of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, rheumatologic, autoimmune, or metabolic disease
4. Receiving any medication that, in the opinion of the Investigator or designee, may pose a risk of compromising tolerance or compliance
5. Are known to or suspected to be currently abusing alcohol or drugs, or have a history (within the past 12 months) of active alcohol or drug abuse
6. Participation in another drug or biologic study within 30 days preceding randomization into this study or during participation in this study
7. Subjects who are unable or unwilling, in the opinion of the Investigator, to comply with all study procedures and cooperate fully with study center staff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-03 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The severity of headache measured with a 4 point scale (The Headache Severity Score (HSS)) | 2 hours after dosing
Absence of headache | 2 hours after dosing

SECONDARY OUTCOMES:
The occurence of any type(s) of adverse events(s) | 0-48 hours after dosing
The severity of headache measured with a 4 point scale (The Headache Severity Score (HSS)) | 0, 1, 2, 4, 8 and 24 hours after dosing
Clinical Disability measured on a 4 point scale | 0, 1, 2, 4, 8 and 24 hours after dosing
Overall evaluation of the study medication | 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Peer Tfelt-Hansen, MD, Dr Med Sci, Principal Investigator — Department of Neurology, Glostrup Hospital, Denmark
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Lassen LH, Christiansen I, Iversen HK, Jansen-Olesen I, Olesen J. The effect of nitric oxide synthase inhibition on histamine induced headache and arterial dilatation in migraineurs. Cephalalgia. 2003 Nov;23(9):877-86. doi: 10.1046/j.1468-2982.2003.00586.x. PMID 14616929
- [Background] Afridi S, Kaube H, Goadsby PJ. Occipital activation in glyceryl trinitrate induced migraine with visual aura. J Neurol Neurosurg Psychiatry. 2005 Aug;76(8):1158-60. doi: 10.1136/jnnp.2004.050633. PMID 16024898
- [Background] Alderton WK, Cooper CE, Knowles RG. Nitric oxide synthases: structure, function and inhibition. Biochem J. 2001 Aug 1;357(Pt 3):593-615. doi: 10.1042/0264-6021:3570593. PMID 11463332
- [Background] Burstein R, Collins B, Jakubowski M. Defeating migraine pain with triptans: a race against the development of cutaneous allodynia. Ann Neurol. 2004 Jan;55(1):19-26. doi: 10.1002/ana.10786. PMID 14705108
- [Background] Costa A, Smeraldi A, Tassorelli C, Greco R, Nappi G. Effects of acute and chronic restraint stress on nitroglycerin-induced hyperalgesia in rats. Neurosci Lett. 2005 Jul 22-29;383(1-2):7-11. doi: 10.1016/j.neulet.2005.03.026. Epub 2005 Apr 18. PMID 15936504
- [Background] Handy RL, Moore PK. Effects of selective inhibitors of neuronal nitric oxide synthase on carrageenan-induced mechanical and thermal hyperalgesia. Neuropharmacology. 1998;37(1):37-43. doi: 10.1016/s0028-3908(97)00201-3. PMID 9680257
- [Background] Heinzen EL, Pollack GM. Pharmacodynamics of morphine-induced neuronal nitric oxide production and antinociceptive tolerance development. Brain Res. 2004 Oct 15;1023(2):175-84. doi: 10.1016/j.brainres.2004.07.015. PMID 15374743
- [Background] Inoue T, Mashimo T, Shibata M, Shibuta S, Yoshiya I. Rapid development of nitric oxide-induced hyperalgesia depends on an alternate to the cGMP-mediated pathway in the rat neuropathic pain model. Brain Res. 1998 May 11;792(2):263-70. doi: 10.1016/s0006-8993(98)00147-4. PMID 9593928
- [Background] Levy D, Zochodne DW. NO pain: potential roles of nitric oxide in neuropathic pain. Pain Pract. 2004 Mar;4(1):11-8. doi: 10.1111/j.1533-2500.2004.04002.x. PMID 17129298
- [Background] Martelletti P, D'Alo S, Stirparo G, Rinaldi C, Cifone MG, Giacovazzo M. Modulation of nitric oxide synthase by nitric oxide donor compounds in migraine. Int J Clin Lab Res. 1998;28(2):135-9. doi: 10.1007/s005990050033. PMID 9689557
- [Background] Mungrue IN, Bredt DS, Stewart DJ, Husain M. From molecules to mammals: what's NOS got to do with it? Acta Physiol Scand. 2003 Oct;179(2):123-35. doi: 10.1046/j.1365-201X.2003.01182.x. PMID 14510775
- [Background] Naik AK, Tandan SK, Kumar D, Dudhgaonkar SP. Nitric oxide and its modulators in chronic constriction injury-induced neuropathic pain in rats. Eur J Pharmacol. 2006 Jan 13;530(1-2):59-69. doi: 10.1016/j.ejphar.2005.11.029. Epub 2005 Dec 20. PMID 16364289
- [Background] Osborne MG, Coderre TJ. Effects of intrathecal administration of nitric oxide synthase inhibitors on carrageenan-induced thermal hyperalgesia. Br J Pharmacol. 1999 Apr;126(8):1840-6. doi: 10.1038/sj.bjp.0702508. PMID 10372828
- [Background] Shimomura T, Murakami F, Kotani K, Ikawa S, Kono S. Platelet nitric oxide metabolites in migraine. Cephalalgia. 1999 May;19(4):218-22. doi: 10.1046/j.1468-2982.1999.019004218.x. PMID 10376166
- [Background] Taffi R, Vignini A, Lanciotti C, Luconi R, Nanetti L, Mazzanti L, Provinciali L, Silvestrini M, Bartolini M. Platelet membrane fluidity and peroxynitrite levels in migraine patients during headache-free periods. Cephalalgia. 2005 May;25(5):353-8. doi: 10.1111/j.1468-2982.2004.00863.x. PMID 15839850
- [Background] Tfelt-Hansen P, De Vries P, Saxena PR. Triptans in migraine: a comparative review of pharmacology, pharmacokinetics and efficacy. Drugs. 2000 Dec;60(6):1259-87. doi: 10.2165/00003495-200060060-00003. PMID 11152011
- [Background] Thomsen LL, Olesen J. Nitric oxide theory of migraine. Clin Neurosci. 1998;5(1):28-33. PMID 9523055
- [Background] van der Kuy PH, Lohman JJ. The role of nitric oxide in vascular headache. Pharm World Sci. 2003 Aug;25(4):146-51. doi: 10.1023/a:1024800512790. PMID 12964492
- [Background] Yoon YW, Sung B, Chung JM. Nitric oxide mediates behavioral signs of neuropathic pain in an experimental rat model. Neuroreport. 1998 Feb 16;9(3):367-72. doi: 10.1097/00001756-199802160-00002. PMID 9512373